CLINICAL TRIAL: NCT04495621
Title: Open-label, Multicentre, Phase Ib/II Study of MEN1611, a PI3K Inhibitor, and Cetuximab in Patients With PIK3CA Mutated Metastatic Colorectal Cancer Failing Irinotecan, Oxaliplatin, 5-FU and Anti-EGFR Containing Regimens
Brief Title: MEN1611 With Cetuximab in Metastatic Colorectal Cancer (C-PRECISE-01)
Acronym: C-PRECISE-01
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Menarini Group (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: MEN1611-02; 2019-003727-38 (EudraCT Number)
Record Dates: First submitted 2020-06-30; First posted 2020-08-03 (Actual); Results first posted 2025-05-01 (Actual); Last update posted 2025-05-01 (Actual); Status verified 2025-04

CONDITIONS: Metastatic Colorectal Cancer
Keywords: Metastatic Colorectal Cancer; PI3K Inhibitor; PIK3CA mutated; MEN1611; Cetuximab; anti-EGFR; mCRC
MeSH Terms: conditions — Colorectal Neoplasms | interventions — Cetuximab

STUDY DESIGN:
Intervention Model Description: Step 1: Confirmation of Dose for Cohort Expansion / Step 2: Cohort Expansion
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- MEN1611 (Experimental): MEN1611 + Cetuximab
  Interventions: Drug: MEN1611; Drug: Cetuximab

INTERVENTIONS:
Drug: MEN1611 — MEN1611 oral dose administered twice daily for a continuous 28-day cycle.
Drug: Cetuximab — Cetuximab solution for infusion administered weekly via intravenous infusion.

SUMMARY:
Open-label, dose-confirmation and cohort expansion, multicenter, Phase Ib/II study to assess the anti-tumor activity and safety of MEN1611 in combination with cetuximab for the treatment of participants with phosphatidylinositol 3-kinase, catalytic, alpha polypeptide gene (PIK3CA)-mutated metastatic colorectal cancer.

DETAILED DESCRIPTION:
This Phase Ib/II study investigated the anti-tumor activity and safety of daily oral doses MEN1611 in combination with cetuximab in female and male participants affected by PIK3CA-mutated, neuroblastoma-Kristen-rat sarcoma virus (N-K-RAS) wild-type, and BRAF wild-type metastatic colorectal cancer.

MEN1611 is a potent, selective class I phosphoinositide 3-kinase (PI3K) inhibitor. The maximum tolerated dose of MEN1611 given as single agent was assessed in a Phase I trial in participants with advanced solid tumors.

This Phase Ib/II started with a dose confirmation part (Step 1) to identify the recommended phase 2 dose of MEN1611 given in combination with cetuximab.

The study continued with a cohort expansion (Step 2) to explore the anti-tumor activity of the selected MEN1611 dose level combined with cetuximab with further assessment of safety and tolerability.

ELIGIBILITY:
Main Inclusion Criteria:

* Histological documentation of adenocarcinoma of the colon or rectum.
* Progression or recurrence following prior irinotecan, oxaliplatin, 5-fluorouracil (5-FU) and anti-epidermal growth factor receptor (EGFR) containing regimens for metastatic disease.
* Best response according to Response Evaluation Criteria in Solid Tumours (RECIST) criteria to the last anti-EGFR containing regimen of partial response or stable disease for at least 4 months.
* Measurable disease according to RECIST criteria.
* N-K-RAS (exons 2, 3 and 4) and BRAF wild-type and PIK3CA mutated.
* Eastern Cooperative Oncology Group performance status of 0 or 1.

Main Exclusion Criteria:

* Previous treatment with PI3K inhibitor.
* Brain metastases, unless treated >4 weeks before screening visit and only if clinically stable and not receiving corticosteroids.
* National Cancer Institute Common Terminology Criteria for Adverse Events v5.0 Grade ≥2 diarrhea.
* History of significant, uncontrolled or active cardiovascular disease.
* Known active or uncontrolled pulmonary dysfunction.
* Uncontrolled diabetes mellitus (glycated hemoglobin >7%) and fasting plasma glucose >126 milligrams/deciliter.
* Known history of human immunodeficiency virus infection or active infection with hepatitis C virus or hepatitis B virus.
* Concurrent chronic immunosuppressive treatment either with steroids or other immunosuppressive agents.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2020-07-20 (Actual); Primary Completion 2024-01-12 (Actual); Study Completion 2024-02-27 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Josep Tabernero, MD, PhD, Study Chair — Vall d' Hebron Institute of Oncology (VHIO), Barcelona, Spain
Locations (28):
- United States (3):
  - Mayo Clinic Arizona, Phoenix, Arizona
  - The Oncology Institute of Hope and Innovation, Anaheim, California
  - MultiCare Health System Institute for Research and Innovation, Tacoma, Washington
- France (3):
  - ICO - Site Paul Papin, Angers
  - Centre Georges François Leclerc, Dijon
  - ICO - Site René Gauducheau, Saint-Herblain
- Germany (6):
  - Charite Universitaetsmedizin Berlin - Campus Benjamin Franklin, Berlin
  - Universitaetsklinikum Carl Gustav Carus TU Dresden, Dresden
  - Asklepios Klinik Altona, Hamburg
  - Klinikum der Universitaet Muenchen Campus Grosshadern, Munich
  - Klinikum rechts der Isar der TU, Munich
  - Universitaetsklinikum Tuebingen, Tübingen
- Italy (5):
  - Azienda Ospedaliero Universitaria San Martino, Genoa
  - Istituto Europeo di Oncologia (IEO), Milan
  - Azienda Socio Sanitaria Territoriale Niguarda, Milan
  - Azienda Ospedaliero Universitaria Pisana, Pisa
  - Istituto Clinico Humanitas, Rozzano
- Netherlands (4):
  - Amsterdam University Medical Center, Amsterdam
  - Maastricht University Medical Center, Maastricht
  - Radboud Nijmegen, Nijmegen
  - Erasmus Medisch Centrum, Rotterdam
- Poland (2):
  - Examen sp. z o.o., Skórzewo
  - Centrum Onkologii-Instytut im.M.Sklodowskiej Curie, Warsaw
- Spain (5):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Hospital Universitario Ramon y Cajal, Madrid
  - Fundacion Jimenez Diaz, Madrid
  - Centro Integral Oncologico Clara Campal, Madrid
  - Hospital Clinico Universitario de Valencia, Valencia

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase 1b (Dose Confirmation); Phase 2 (Cohort Expansion): Participants received MEN1611 twice daily and cetuximab weekly, every 28-day cycle.
Period: Overall Study
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
Started | 7 | 22
Received At Least 1 Dose of Study Drug (Safety Population) | 7 | 22
Completed | 0 | 0
Not Completed | 7 | 22
Not completed — Withdrawal by Subject | 0 | 3
Not completed — Death | 7 | 11
Not completed — Investigator Decision | 0 | 7
Not completed — Lost to Follow-up | 0 | 1

BASELINE CHARACTERISTICS:
Population: Safety Population: all participants who received at least 1 dose of MEN1611.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion) | Total
Number analyzed (Participants) | 7 | 22 | 29
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.9 (12.16) | 58.9 (12.38) | 57.7 (12.31)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 11 | 12
  Male | 6 | 11 | 17
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0
  Not Hispanic or Latino | 7 | 15 | 22
  Unknown or Not Reported | 0 | 7 | 7

OUTCOME MEASURES:

1. Primary Outcome: Phase 1b: Recommended Phase 2 Dose (RP2D) of MEN1611 in Combination With Cetuximab
Description: RP2D was defined as the highest dose level in milligrams (mg) at which no more than 1 participant during the dose confirmation phase (Phase 1b) experienced a dose-limiting toxicity (DLT) during the DLT assessment window (28 days), or the maximum dose judged to be tolerable by the data safety committee.
Time Frame: Day 1 through Day 28 of Cycle 1 (28 days/cycle)
Population: Safety Population: all participants who received at least 1 dose of MEN1611. As pre-specified, RP2D data were collected and are reported for 'Phase 1b (Dose Confirmation)' cohort only.
Measure: Number; unit: mg
Arm/Group | Phase 1b (Dose Confirmation)
Number analyzed (Participants) | 7
mg | 48

2. Primary Outcome: Best Overall Response Rate (ORR) of MEN1611 in Combination With Cetuximab
Description: The best ORR was defined as percentage of participants who had a best overall response to therapy of complete response (CR), partial response (PR), stable disease (SD), or progressive disease (PD) and was defined according to Response Evaluation Criteria in Solid Tumors version 1.1 assessment locally performed using computed tomography scans or magnetic resonance imaging of the chest and abdomen (including pelvis and adrenal glands).
Time Frame: Up to 37 Months
Population: Efficacy Population: all participants who received at least 2 complete treatment cycles and had at least 1 disease assessment.
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
Number analyzed (Participants) | 5 | 14
percentage of participants
  Complete Response | 0.0 | 7.1
  Partial Response | 40.0 | 7.1
  Stable Disease | 40.0 | 57.1
  Progressive Disease | 20.0 | 28.6

3. Primary Outcome: Phase 1b: Number of Participants With DLTs for MEN1611
Description: A DLT was defined as any of the following adverse drug reactions (ADRs) related to the combination regimens or to MEN1611 alone and unrelated to the participants' underlying disease or concomitant medication occurring during Cycle 1 over the DLT assessment window of 28 days: any Grade 3 (lasting >7 days) or Grade 4 increase in aspartate aminotransferase, alanine aminotransferase, or alkaline phosphatase; any Grade ≥3 cardiac disorder or new segmental wall-motion abnormalities; any Grade ≥3 non-hematologic toxicity with the following exceptions: nausea, vomiting, diarrhea, skin rash, hyperglycemia. An ADR was defined as any adverse event suspected by the investigator and/or the sponsor to be related to MEN1611, cetuximab, or both given in combination.
Time Frame: Day 1 through Day 28 of Cycle 1 (28 days/cycle)
Population: Dose-limiting Toxicity (DLT) Population: all participants who received at least 80% of MEN1611 and 75% of cetuximab during Cycle 1 with a safety follow-up of 28 days after the first administration of the study treatment. Any participant who experienced DLT was also considered evaluable, regardless of the dose received. As pre-specified, data were collected and reported for the 'Phase 1b (Dose Confirmation)' cohort only.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase 1b (Dose Confirmation)
Number analyzed (Participants) | 6
Participants | 0

4. Secondary Outcome: Plasma Concentration of MEN1611 in Combination With Cetuximab
Description: Blood samples were taken for the analyses of MEN1611 in plasma at designated time points. Results are reported as nanograms/millilitre (ng/mL).
Time Frame: Day 22 (1.5 hours postdose) of Cycle 1 (28 days/cycle)
Population: Pharmacokinetics (PK) Set: all participants who received MEN1611 and for whom a PK sample was obtained and analyzed. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
Number analyzed (Participants) | 7 | 1
ng/mL | 173.37 (125.513) | 241.2 (NA) — Standard deviation is not calculable for 1 participant.

5. Secondary Outcome: Disease Control Rate (DCR) of MEN1611 in Combination With Cetuximab
Description: DCR was defined as percentage of participants whose disease shrank or remained stable over a certain time period and was calculated based on the sum of the CR, PR, and SD rates according to local assessment.
Time Frame: Up to 37 Months
Population: as for outcome 2
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
Number analyzed (Participants) | 5 | 14
percentage of participants | 80 [28.4 to 99.5] | 71.4 [41.9 to 91.6]

6. Secondary Outcome: Duration of Response (DOR) of MEN1611 in Combination With Cetuximab
Description: DOR was defined as the time from confirmation of a PR, CR or SD as locally assessed, until the disease had been shown to progress following treatment. Participants with a previous response who did not show a relapse or died without recording a relapse were censored at their last available relapse-free tumor assessment date. Participants with only one tumor assessment after baseline showing a PD were not included in the calculation.
Time Frame: Up to 37 months
Population: Efficacy Population: all participants who received at least 2 complete treatment cycles and had at least 1 disease assessment. Here, 'Overall Number of Participants Analyzed' signifies those participants who were evaluable for this outcome measure.
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
Number analyzed (Participants) | 4 | 10
days | 85 [47 to NA] — Values were non-estimable (insufficient number of participants with events). | 169 [120 to NA] — Values were non-estimable (insufficient number of participants with events).

7. Secondary Outcome: Progression-free Survival (PFS) of MEN1611 in Combination With Cetuximab
Description: PFS was defined as the number of days between the first study treatment administration to the date of first documented disease progression as per local assessment, relapse or death from any cause. Responding participants and participants who were lost to follow-up were censored at their last tumor assessment date.
Time Frame: Up to 37 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
Number analyzed (Participants) | 5 | 14
days | 121 [75 to NA] — Values were non-estimable (insufficient number of participants with events). | 162 [57 to 218]

8. Secondary Outcome: Overall Survival (OS) of MEN1611 in Combination With Cetuximab
Description: OS was defined as the number of days between the first study treatment administration and death from any cause. Participants still alive that had withdrawn from the study were censored using the latest among end of study and follow-up dates. Drop-out participants were considered censored and the last available date in which the participant was known to be alive was considered.
Time Frame: Up to 37 months
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
Number analyzed (Participants) | 5 | 14
days | 471 [171 to NA] — Values were non-estimable (insufficient number of participants with events). | 308 [177 to NA] — Values were non-estimable (insufficient number of participants with events).

ADVERSE EVENTS:
Time Frame: From Day 1 to the end of study (37 months)
Description: All reported safety data based upon the Safety Population: all participants who received at least 1 dose of MEN1611.
Arm/Group | Phase 1b (Dose Confirmation) | Phase 2 (Cohort Expansion)
All-Cause Mortality (participants affected / at risk) | 7/7 | 11/22
Serious Adverse Events (participants affected / at risk) | 5/7 | 11/22
Other Adverse Events (participants affected / at risk) | 7/7 | 22/22
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1b (Dose Confirmation) (N=7) | Phase 2 (Cohort Expansion) (N=22)
Hypotension (Vascular disorders) | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 1
Asthenia (General disorders) | 0 | 1
Pyrexia (General disorders) | 0 | 1
Abdominal pain (Gastrointestinal disorders) | 0 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Diarrhoea (Gastrointestinal disorders) | 0 | 1
Enterovesical fistula (Gastrointestinal disorders) | 1 | 0
Gastrointestinal necrosis (Gastrointestinal disorders) | 0 | 1
Intestinal obstruction (Gastrointestinal disorders) | 0 | 1
Cholangitis (Hepatobiliary disorders) | 0 | 2
Jaundice cholestatic (Hepatobiliary disorders) | 0 | 1
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 1 | 0
Fistula (Musculoskeletal and connective tissue disorders) | 0 | 1
Anal abscess (Infections and infestations) | 0 | 1
Biliary tract infection (Infections and infestations) | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0
Influenza (Infections and infestations) | 0 | 1
Sepsis (Infections and infestations) | 0 | 1
Staphylococcal infection (Infections and infestations) | 0 | 1
Decreased appetite (Metabolism and nutrition disorders) | 0 | 1
Hyperglycaemia (Metabolism and nutrition disorders) | 1 | 1
Hypernatraemia (Metabolism and nutrition disorders) | 0 | 1
Hypomagnesaemia (Metabolism and nutrition disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk, or affected / at risk where a term's number at risk differs:
Term (organ system) | Phase 1b (Dose Confirmation) (N=7) | Phase 2 (Cohort Expansion) (N=22)
Asthenia (General disorders) | 0 | 9
Chills (General disorders) | 0 | 2
Condition aggravated (General disorders) | 1 | 0
Fatigue (General disorders) | 3 | 1
Mucosal inflammation (General disorders) | 0 | 7
Oedema peripheral (General disorders) | 2 | 1
Pyrexia (General disorders) | 2 | 6
Vaccination site pain (General disorders) | 1 | 0
Xerosis (General disorders) | 0 | 2
Scrotal swelling (Reproductive system and breast disorders) | 1/6 | 0/11 — This adverse event affected only male participants.
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 2
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 3
Alanine aminotransferase increased (Investigations) | 0 | 2
Amylase increased (Investigations) | 1 | 1
Aspartate aminotransferase increased (Investigations) | 1 | 2
Blood albumin decreased (Investigations) | 0 | 2
Blood alkaline phosphatase increased (Investigations) | 1 | 0
Blood lactate dehydrogenase increased (Investigations) | 0 | 2
Blood potassium decreased (Investigations) | 0 | 3
Blood pressure increased (Investigations) | 1 | 0
Blood uric acid increased (Investigations) | 0 | 2
Gamma-glutamyltransferase increased (Investigations) | 1 | 1
Lipase increased (Investigations) | 1 | 1
Platelet count decreased (Investigations) | 0 | 2
Protein total decreased (Investigations) | 0 | 2
SARS-CoV-2 test positive (Investigations) | 1 | 0
Transaminases increased (Investigations) | 0 | 2
Weight decreased (Investigations) | 2 | 5
Sinus tachycardia (Cardiac disorders) | 1 | 0
Supraventricular tachycardia (Cardiac disorders) | 1 | 0
Dizziness (Nervous system disorders) | 1 | 1
Dysgeusia (Nervous system disorders) | 1 | 2
Headache (Nervous system disorders) | 0 | 3
Neuropathy peripheral (Nervous system disorders) | 1 | 0
Neurotoxicity (Nervous system disorders) | 0 | 2
Anaemia (Blood and lymphatic system disorders) | 4 | 6
Lymphopenia (Blood and lymphatic system disorders) | 1 | 2
Abdominal pain (Gastrointestinal disorders) | 0 | 3
Diarrhoea (Gastrointestinal disorders) | 5 | 16
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 0 | 2
Nausea (Gastrointestinal disorders) | 1 | 7
Stomatitis (Gastrointestinal disorders) | 2 | 2
Vomiting (Gastrointestinal disorders) | 0 | 5
Dyspepsia (Gastrointestinal disorders) | 1 | 2
Hepatic cytolysis (Hepatobiliary disorders) | 0 | 2
Hyperbilirubinaemia (Hepatobiliary disorders) | 1 | 1
Alopecia (Skin and subcutaneous tissue disorders) | 0 | 2
Decubitus ulcer (Skin and subcutaneous tissue disorders) | 1 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 5
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 3
Eczema (Skin and subcutaneous tissue disorders) | 0 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 2
Palmar erythema (Skin and subcutaneous tissue disorders) | 1 | 0
Palmar-plantar erythrodysaesthesia syndrome (Skin and subcutaneous tissue disorders) | 0 | 5
Pruritus (Skin and subcutaneous tissue disorders) | 1 | 3
Rash (Skin and subcutaneous tissue disorders) | 7 | 11
Skin fissures (Skin and subcutaneous tissue disorders) | 0 | 3
Skin toxicity (Skin and subcutaneous tissue disorders) | 0 | 3
Acute kidney injury (Renal and urinary disorders) | 0 | 2
Haematuria (Renal and urinary disorders) | 1 | 0
Myalgia (Musculoskeletal and connective tissue disorders) | 0 | 2
Clostridium difficile infection (Infections and infestations) | 1 | 0
Conjunctivitis (Infections and infestations) | 0 | 4
COVID-19 (Infections and infestations) | 0 | 3
Escherichia infection (Infections and infestations) | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 1 | 0
Folliculitis (Infections and infestations) | 0 | 3
Localised infection (Infections and infestations) | 1 | 0
Oral herpes (Infections and infestations) | 1 | 0
Paronychia (Infections and infestations) | 3 | 5
Staphylococcal infection (Infections and infestations) | 1 | 0
Upper respiratory tract infection (Infections and infestations) | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 7
Hyperglycaemia (Metabolism and nutrition disorders) | 3 | 13
Hypoalbuminaemia (Metabolism and nutrition disorders) | 1 | 1
Hypocalcaemia (Metabolism and nutrition disorders) | 2 | 1
Hypokalaemia (Metabolism and nutrition disorders) | 2 | 2
Hypomagnesaemia (Metabolism and nutrition disorders) | 3 | 8
Hypophosphataemia (Metabolism and nutrition disorders) | 2 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The results of the study cannot be submitted for presentation, abstract, poster exhibition, or publication by the investigator until Menarini Ricerche S.p.A. has reviewed/commented and agreed to any publication.

DOCUMENTS (2):
  • Study Protocol (2023-05-15): https://cdn.clinicaltrials.gov/large-docs/21/NCT04495621/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-11): https://cdn.clinicaltrials.gov/large-docs/21/NCT04495621/SAP_001.pdf